CLINICAL TRIAL: NCT00930436
Title: Evaluation of Sodium Bicarbonate to Reduce Chronic Kidney Injury in Subjects With Advanced Chronic Kidney Disease (CKD) Who Are Undergoing Angiography
Brief Title: Evaluation of Sodium Bicarbonate to Reduce the Incidence of Contrast Induced Chronic Kidney Injury in Patients With Kidney Disease
Acronym: BOSS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: MD Scientific (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MDS001
Record Dates: First submitted 2009-06-26; First posted 2009-06-30 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-02

CONDITIONS: Contrast Induced Kidney Injury.
Keywords: chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline infusion (Active Comparator): Saline will be given as an active control agent to compare with sodium bicarbonate. Each bag of solution will be blinded, and given in the same manner.
  Interventions: Drug: sodium bicarbonate
- Sodium Bicarbonate (Experimental): Infusion of sodium bicarbonate will be given prior to,during and after the contrast agent for a total of 6 to 10 hours
  Interventions: Drug: sodium bicarbonate

INTERVENTIONS:
Drug: sodium bicarbonate — Serum creatinine will be measured on Days 3,7, 30, 90, and 180

SUMMARY:
Patients with Stage 3B, 4,or 5 Chronic Kidney Disease who are to undergo an angiography procedure with contrast agent will be asked if they are willing to join the trial. If so they will be screened and randomized to receive either sodium bicarbonate or saline before, during and after the contrast media is given. They will be asked for serum samples 1 to 3 days, 7, 30, 90 and 180 days after the procedure to evaluate whether the sodium bicarbonate has reduced the incidence of contrast induced chronic kidney disease by measuring their serum creatinine, as well as whether they have required renal dialysis or other renal replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for angiography
* Stage 3B, 4 or 5 Chronic kidney disease (i.e. eGFR <=44)
* Either sex over 18 years of age

Exclusion Criteria:

* Pregnant or breast feeding
* On any kidney replacement list
* Gastric tube in place or gastric drainage
* Uncorrected hypoglycemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2010-01; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Death or renal replacement therapy or sustained kidney injury | Over six months following treatment
  Sustained kidney injury is two sequential 20% reduction of eGFR from baseline as calculated from change in sertum creatinine at least three weeks after receiving IP.

SECONDARY OUTCOMES:
A comparison between the treatments for length of hospital stay, post contrast. | Over six months after the treatment
A comparison between the treatments of the time to renal replacement therapy (any type) or death (whichever occurs first) over the 6-month observation period. | six months after receiving IP

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Osceola Regional Medical Center, Kissimmee, Florida
  - Northside Hospital, St. Petersburg, Florida
  - Redmond Regional Medical Center, Rome, Georgia
  - St. Johns Hospital, Springfield, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - St Luke's Health System, Kansas City, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mt Sinai School of Medcine, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - The Christ Hospital, Cincinnati, Ohio
  - St Luke's Heart and Vascular Center, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital (Lifespan), Providence, Rhode Island
  - Centennial Medical Center, Nashville, Tennessee
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - Fletcher Allen Hospital, Burlington, Vermont